CLINICAL TRIAL: NCT05030441
Title: A Pilot Study of Ivosidenib for Patients With Clonal Cytopenia of Undetermined Significance and Mutations in IDH1
Brief Title: Ivosidenib for Patients With Clonal Cytopenia of Undetermined Significance and Mutations in IDH1
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Servier Hellas Pharmaceuticals Ltd. (Industry); Gateway for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202110038
Record Dates: First submitted 2021-08-24; First posted 2021-09-01 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Clonal Cytopenia of Undetermined Significance
MeSH Terms: interventions — ivosidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ivosidenib (Experimental): -Ivosidenib is an oral drug which will be administered on an outpatient basis at a dose of 500 mg daily for up to 5 years. Each cycle is 28 days.
  Interventions: Drug: Ivosidenib

INTERVENTIONS:
Drug: Ivosidenib — . Patients should take ivosidenib at approximately the same time every day, with or without food, but should be instructed to avoid a high-fat meal as well as grapefruit and grapefruit products.
  Other Names: TIBSOVO

SUMMARY:
This is an open-label, multicenter study exploring the efficacy of ivosidenib in patients with clonal cytopenia of undetermined significance (CCUS) with mutations in IDH1. The purpose is to establish proof of principle that ivosidenib is well-tolerated and potentially efficacious in improving blood count abnormalities in these patients.

The study will also be offered in a decentralized, remote structure to patients.

ELIGIBILITY:
Inclusion Criteria:

* Unexplained cytopenia for at least 6 months. Cytopenia is defined as the presence of ≥1 blood count indexes below the following thresholds:

  * Hgb <10 g/dL
  * ANC <1.8 × 10^9/L
  * Platelets <100 × 10^9/L
* IDH1 gene mutation (R132) confirmed by droplet digital PCR (ddPCR) testing, at a frequency > 2%. This will be performed locally and confirmed at Washington University.
* At least 18 years of age.
* ECOG performance status 0-2
* Adequate organ function as defined below:

  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Serum total bilirubin < 1.5 x IULN (an upper limit of bilirubin 5mg/dL is acceptable if it can be attributed to Gilbert's syndrome or erythropoiesis)
  * Serum creatinine < 2 x IULN or creatinine clearance > 50 mL/min by Cockcroft-Gault glomerular filtration rate estimation
* The effects of ivosidenib on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (defined in Section 5.5) prior to study entry, for the duration of study participation, and for 90 days after the last dose of ivosidenib. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of the study, and for 90 days after the last dose of ivosidenib.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Indication of hematologic disease by bone marrow biopsy within 6 months of study entry.

  *Evidence of disease progression from time of bone marrow biopsy to enrollment based on investigator review of symptoms and complete blood counts
* Active malignancy (defined as > 1 cm disease on most recent CT scan in the past 6 months).
* Currently receiving therapy for solid tumor malignancy.
* Currently receiving any other investigational agents.
* Known dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to ivosidenib or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 72 hours of study entry.
* Heartrate corrected QT interval (QTc) > 450 msec or with other factors that increase the risk of QT prolongation or arrhythmic events (e.g. heart failure, hypokalemia, family history of long QT interval syndrome).
* Known medical history of progressive multifocal leukoencephalopathy (PML).
* Currently taking medications known to be CYP3A4 strong inducers and sensitive substrates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Rate of improvement in hematologic parameters | Through 30 days after completion of treatment (estimated to be 61 months)
  Will be evaluated according to a modified version of the IWG 2006 Criteria for Hematologic Improvement for patients with MDS on clinical trials
  * Erythroid response (pretreatment, <11 g/DL)
    * Hemoglobin (Hgb) increase by ≥1.5 g/dL
    * Relevant reduction of units of RBC transfusions by an absolute number of at least 4 RBC transfusions/8 weeks, compared with the pretreatment transfusion number in the previous 8 weeks. Only RBC transfusions given for an Hgb of ≤9.0 g/dL pretreatment will count in the RBC transfusion response evaluation
  * Platelet response (pretreatment, <100 x 10^9/L)
    * Absolute increase of ≥30 × 10^9/L for patients starting with >20 × 10^9/L platelets.
    * Increase from <20 × 10^9/L to >20 × 10^9/L and by at least 100%.
  * Neutrophil response (pretreatment, <1.0 x 10^9/L):
    * At least 100% increase and an absolute increase >0.5 × 10^9/L. If pegfilgrastim being used prior to initiation of study, define response as no longer requiring pegfilgrastim to maintain ANC >500.

SECONDARY OUTCOMES:
Change in mutant IDH1 variant allele fraction | Through completion of treatment (estimated to be 60 months)
  -ddPCR is a highly sensitive and accurate method for quantifying VAF. This will be performed centrally at the Washington University clinical pathology laboratory using standard procedures. To account for assay variation, the investigators will perform 10 runs using the ddPCR assay and take the mean VAF as the final measurement.
Disease free survival | Through 30 days after completion of treatment (estimated to be 61 months)
  -Events include development of MDS/AML or death.
Number of adverse events as measured by CTCAE v 5.0 | Through 30 days after completion of treatment (estimated to be 61 months)
Duration of hematologic response | Through completion of treatment (estimated to be 60 months)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Bolton, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - Cleveland Clinic - Case Comprehensive Cancer Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Individual participate data that underlie the results reported in this article after deidentification (including text, tables, figures and appendices) will be available.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will be available immediately following publication with no end date.
Access Criteria: The data will be available immediately following publication with no end date. Access will be provided to anyone and for any purpose.

REFERENCES:
- See also: Preventing IDH Mutant Myeloid Neoplasm (PIMM) Clinical Trial Information — https://sites.wustl.edu/pimm/
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu